CLINICAL TRIAL: NCT01260922
Title: A Relative Bioavailability Study of 10 mg Donepezil Hydrochloride Orally Disintegrating Tablets Under Fasting Conditions.
Brief Title: 10 mg Donepezil Hydrochloride Orally Disintegrating Tablets Under Fasting Conditions.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Responsible Party: Associate Director, Biopharmaceutics, TEVA Pharmaceuticals, USA
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: R05-1254
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Results first posted 2011-02-21 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-01

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational Test Product (Experimental): Donepezil Hydrochloride 10 mg Orally Disintegrating Tablets
  Interventions: Drug: Donepezil Hydrochloride
- Reference Listed Drug (Active Comparator): Aricept® 10 mg Orally Disintegrating Tablets
  Interventions: Drug: Aricept®

INTERVENTIONS:
Drug: Donepezil Hydrochloride — 10 mg Orally Disintegrating Tablet
  Arms: Investigational Test Product
Drug: Aricept® — 10 mg Orally Disintegrating Tablet
  Other Names: Donepezil Hydrochloride (generic name)
  Arms: Reference Listed Drug

SUMMARY:
This study investigated the relative bioavailability (rate and extent of absorption) of Donepezil Hydrochloride Orally Disintegrating Tablets, 10 mg by Teva Pharmaceuticals, USA with that of Aricept® Orally Disintegrating Tablets, Manufactured and Marketed by Eisai Inc., following a single oral dose (1 x 10 mg orally disintegrating tablet) in healthy adult subjects administered under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Screening Demographics: All volunteers for this study will be healthy men and women 18 years of age or older at the time of dosing. The weight range will not exceed + 20% for height and body frame as per Desirable Weights for Adults-1983 Metropolitan Height and Weight Table.
* Screening Procedures: Each volunteer will complete the screening process within 28 days prior to Period I dosing. Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed, and signed by each potential participant before full implementation of screening procedures.
* If female and:

  * of childbearing potential, is practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s); or
  * is postmenopausal for at least 1 year; or
  * is surgically sterile.

Exclusion Criteria:

* Volunteers with a recent history of drug or alcohol addiction or abuse.
* Volunteers with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the clinical investigators).
* Volunteers whose clinical laboratory test values are outside the accepted reference range and when confirmed on reexamination are deemed to be clinically significant.
* Volunteers demonstrating a reactive screen for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody.
* Volunteers demonstrating a positive drug abuse screen when screened for this study.
* Female volunteers demonstrating a positive pregnancy screen.
* Female volunteers who are currently breastfeeding.
* Volunteers with a history of allergic response(s) to donepezil or related drugs.
* Volunteers with a history of clinically significant allergies including drug allergies.
* Volunteers with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigators).
* Volunteers who currently use tobacco products.
* Volunteers who have taken any drug known to induce or inhibit hepatic drug metabolism in the 28 days prior to Period I dosing.
* Volunteers who report donating greater than 150 mL of blood within the 28 days prior to Period I dosing.
* Volunteers who have donated plasma within 14 days prior to Period I dosing.
* Volunteers who report receiving any investigational drug within 28 days prior to Period I dosing.
* Volunteers who report taking any systemic prescription medication in the 14 days prior to Period I dosing.
* Female volunteers who report the use of oral contraceptives or injectable contraceptives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-04; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Carlson, Pharm.D., Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., East Grand Forks, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Donepezil Hydrochloride (Test) First: 10 mg Donepezil Hydrochloride Orally Disintegrating Tablets test product dosed in first period followed by 10 mg Aricept® Orally Disintegrating Tablets reference product dosed in the second period.
- Aricept® (Reference) First: 10 mg Aricept® Orally Disintegrating Tablets reference product dosed in first period followed by 10 mg Donepezil Hydrochloride Orally Disintegrating Tablets test product dosed in the second period.
Period: First Intervention
Arm/Group | Donepezil Hydrochloride (Test) First | Aricept® (Reference) First
Started | 13 | 13
Completed | 13 | 12
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout of 28 Days
Arm/Group | Donepezil Hydrochloride (Test) First | Aricept® (Reference) First
Started | 13 | 12
Completed | 9 | 10
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 4 | 2
Period: Second Intervention
Arm/Group | Donepezil Hydrochloride (Test) First | Aricept® (Reference) First
Started | 9 | 10
Completed | 9 | 8
Not Completed | 0 | 2
Not completed — Emesis | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donepezil Hydrochloride (Test) First | Aricept® (Reference) First | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 6 | 4 | 10
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 1 | 0 | 1
  Caucasian | 12 | 13 | 25
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Donepezil.
Description: Bioequivalence based on Donepezil Cmax (maximum observed concentration of drug substance in plasma).
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Donepezil Hydrochloride (Test): 10 mg Donepezil Hydrochloride Orally Disintegrating Tablets test product dosed in either period.
- Aricept® (Reference): 10 mg Aricept® Orally Disintegrating Tablets reference product dosed in either period.
Arm/Group | Donepezil Hydrochloride (Test) | Aricept® (Reference)
Number analyzed (Participants) | 17 | 17
ng/mL | 17800.27 (4515.36) | 17280.23 (4032.57)
Statistical Analysis 1: Comparison: Donepezil Hydrochloride (Test) vs Aricept® (Reference); Test type: Non-Inferiority or Equivalence — ANOVA is to be used to identify the source contributions by factors including subjects, period, formulation and potential interactions. The geometric mean ratio together with the ANOVA residual mean error term are used to identify the statistical basis for the 90% confidence interval for the ratio of the population means (Test [T]/Reference[R]) of the identified metrics (e.g. AUC, Cmax); Ratio of the T/R geometric mean x 100 = 102.16, 90% CI 2-sided [97.07 to 107.51] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference (R) and test (T) product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t of Donepezil.
Description: Bioequivalence based on Donepezil AUC0-t (area under the concentration-time curve from time zero to time of last measurable concentration).
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Donepezil Hydrochloride (Test) | Aricept® (Reference)
Number analyzed (Participants) | 17 | 17
ng*h/mL | 466307.49 (85094.55) | 490716.21 (86199.11)
Statistical Analysis 1: Comparison: Donepezil Hydrochloride (Test) vs Aricept® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Slope = 94.75, 90% CI 2-sided [92.11 to 97.46] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study, which was approximately 8 weeks in duration.
Description: Volunteers were monitored throughout the study for any adverse experiences. AEs were collected through both solicited and unsolicited methods. The volunteers were encouraged to report signs, symptoms, and any changes in health to the clinic staff.
Arm/Group | Donepezil Hydrochloride (Test) First | Aricept® (Reference) First
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 10/26 | 6/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil Hydrochloride (Test) First (N=26) | Aricept® (Reference) First (N=26)
Headache (General disorders) | 3 (3) | 1 (1)
Nausea (General disorders) | 5 (5) | 4 (5)
Vomiting (General disorders) | 5 (13) | 3 (4)
Dizziness (General disorders) | 0 (0) | 2 (2)
Abnormal Dreams (General disorders) | 2 (2) | 0 (0)
Feeling Hot (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.